CLINICAL TRIAL: NCT01004692
Title: The Effect of Occlusal Splints on Sleep and Respiratory Variables of OSA Patients
Brief Title: The Effect of Occlusal Splints on Respiratory Variables in Obstructive Sleep Apnea (OSA) Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Maria Nikolopoulou, ACTA
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL23988.048.08; METC 0832
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Occlusal splints — The splint will be a hard acrylic-resin stabilization appliance to wear in the upper jaw. The OSS does not come in contact with the gums of the patient and does not act as an orthodontic device. The OSS will be used only for the three nights in a row, of the ambulatory-PSG recording with the OSS in situ.
  Other Names: occlusal stabilisation splint

SUMMARY:
Rationale: The effect of vertical dimension on sleep apnoea and respiratory variables in obstructive sleep apnoea patients.

Objective: To what extend should a possible worsening of the OSA condition, caused by an increase of mouth opening be taken into consideration in daily dental practice, when an occlusal stabilization splint (OSS) is placed in the mouth.

Study design: Cross over RCT-design Study population: OSA patients referred to ACTA from the Slotervaart Hospital, for treatment with a Mandibular Advancement Device (MAD), at least 18 years old.

Intervention: Occlusal stabilization splint (OSS) for the upper jaw and a controlled condition in a cross-over design Main study parameters/endpoints: Apnoea- Hypopnoea Index (AHI) and the Epworth Sleepiness Scale (ESS).

The aim of this study is to determine the effect of vertical dimension of OS on sleep and respiratory variables in OSA patients. The hypothesis is that insertion of an OSS and an increase of the vertical dimension will result in a significant increase in the AHI.

DETAILED DESCRIPTION:
Mild or Moderate OSA patients (AHI 10-30) referred by Slotervaart Hospital, to ACTA, for treatment with an MAD. Both males and females will participate in the study. All participants will be over 18 years old.

Inclusion criteria

* All patients invited should be at least 18 years old.
* OSA patients, diagnosis based on a baseline polysomnographic recording (at the hospital) with AHI values until 30 (mild+ moderate OSAS).
* Adequate retention in the dentition for an occlusal stabilization splint (OSS).

Exclusion criteria

* Medicine usage that influence sleep (eg Benzodiazepines).
* BMI more than 40
* Unhealthy dentition.
* Severe bruxers
* TMD patients An occlusal stabilization splint (OSS) will be constructed for each patient, as an intervention device. The splint will be a hard acrylic-resin stabilization appliance to wear in the upper jaw. The OSS does not come in contact with the gums of the patient and does not act as an orthodontic device. The OSS will be used only for the three nights in a row, of the ambulatory-PSG recording with the OSS in situ.

After written informed consent will be obtained, the patients will be randomly allocated to one of the two groups. To ensure that the groups would be of approx. the same size, block randomization will be used. Block sizes will be used and sizes will vary randomly. The allocation sequence will automatically be generated and subsequently concealed by an independent co-worker, who will keep a paper copy in a lockable drawer.

All patients will be referred to ACTA, by the Center for sleep wake disorders at Slotervaart Hospital. There they will have done a PSG-sleep study. The PSG recording will take place in a dark hospital room, in the Slotervaart Hospital in Amsterdam, at the department of Clinical Neurophysiology (The multidisciplinary Centre for Sleep-Wake Disorders). OSA patients with diagnosis mild and moderate OSA will be invited to participate in the trial.

Following the PSG recording and the diagnosis at Slotervaart Hospital, each patient will come for a first appointment, at the department of Oral Function, section of Oral Kinesiology, at ACTA. Medical and dental history will be obtained. If the patients fulfill the inclusion criteria and agree to participate in the study, impressions of the upper and lower jaw, Body Mass Index (BMI), neck circumference, and the Epworth Sleepiness Scale will be obtained.

The medical history will be obtained by using questionnaires, the dental history by using questionnaires, clinical dental examination, and OPG x-ray (orthopantomogram). The BMI will be obtained by measuring the height and the weight of the patient. (BMI = kg/ cm ²). The neck circumference will be measured in cm. Impressions with alginate and a wax-index with dental wax will be taken for every patient, in order to make the dental casts for the construction of the splints. The whole procedure will last approximately 1 hour.

The patients will be randomly divided in two groups. The patients will be randomly placed in the two groups. The patients will undergo the PSG-recordings without the OSS in situ and the nights with the OSS in situ, in a cross-over design.

Group 1: The patients will undergo 3 nights of home-PSG recording without the OSS in situ first. 2 weeks later they will undergo 3 nights of PSG-recording with the OSS in situ.

Group 2: The patients in Group 2 will first undergo 3 nights of ambulatory PSG-recording with the OSS in situ. 2 weeks later they will undergo 3 nights of home-PSG recording without the OSS in situ.

Appointments will be made either for the OSS placement at ACTA or for the mounting of the equipment for the ambulatory recording, at Slotervaart hospital, depending on in which group the patient will be randomly placed.

Group 1: The mounting of the equipment for the ambulatory recording will take place at the department of Clinical Neurophysiology at Slotervaart Hospital. The procedure will last approximately 1 hour. The Monet hardware (Medcare, Amsterdam, The Netherlands) with 19 recording channels will be used for the recordings and the Rembrandt software will be used for the analysis.

The patient will sleep at home with the ambulatory PSG equipment 3 nights in a row, without the OSS in situ. That means that 3 mounting appointments will be held at the department of Clinical Neurophysiology at Slotervaart Hospital, 3 afternoons in a row.

Every morning after the home PSG-recording, the patients will take off the electrodes themselves at home (using a solution that we will provide them with, in order to resolve the glue) and they will have to bring the equipment back to ACTA.

In the meantime (between the first and the second visit to ACTA), an OSS for the upper jaw will be constructed for every patient. The OSS will be constructed at the same dental laboratory for all patients. It will be made by hard acrylic resin and no palatal coverage will be made.

The patients will come back to ACTA after 1 week (second appointment) for the placement of the splint (OSS). On the second appointment at ACTA the OSS will be placed.

The patients will wear the OSS, in order to get used to it, under the period of one week and after that they will undergo 3 nights of ambulatory sleep recording with the OSS in situ.

Group 2: The patients will come back to ACTA after 1 week (second appointment at ACTA) for the placement of the splint (OSS).

The patients will wear the OSS, in order to get used to it, under the period of one week and after that they will undergo 3 nights of ambulatory sleep recording with the OSS in situ.

The mounting of the equipment for the ambulatory recording will take place at the department of Clinical Neurophysiology at Slotervaart Hospital. The procedure will last approximately 1 hour. The Monet hardware (Medcare, Amsterdam, The Netherlands) with 19 recording channels will be used for the recordings and the Rembrandt software will be used for the analysis.

The patients will sleep at home with the ambulatory PSG equipment 3 days in a row, with the OSS in situ. That means that 3 mounting appointments will be held at the department of Clinical Neurophysiology at Slotervaart Hospital, 3 afternoons in a row.

Every morning after the home PSG-recording, the patients will take off the electrodes themselves at home (using a solution that we will provide them with, in order to resolve the glue) and they will have to bring the equipment back to ACTA.

Two weeks later, the patients that belong in the 2nd group, will undergo 3 ambulatory recordings at home, without the OSS in situ.

All patients will have to fill in 10 questionnaires at the beginning of the study and at the end of the study. The ESS and the "morning- questionnaire" and the evening- questionnaire" will be filled by all patients between nights as well. That means in the beginning, at the end of the study and in the 6 days while having the home- PSG recordings.

Following the last home PSG recording the below mentioned data will be collected (for all patients, belonging to both groups):

* Body Mass Index (BMI)
* Neck circumference
* The Epworth Sleepiness Scale
* Side effects of the splints (OSS).

The main study parameter/ endpoint is the Apnoea-Hypopnoea Index (AHI) value. The secondary study parameter is the Epworth Sleepiness Scale (ESS).

The side effects of the splint (OSS) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* - All patients invited should be at least 18 years old.
* OSA patients, diagnosis based on a baseline polysomnographic recording (at the hospital) with AHI values until 30 (mild+ moderate OSAS).
* Adequate retention in the dentition for an occlusal stabilization splint (OSS).

Exclusion Criteria:

* - Medicine usage that influence sleep (eg Benzodiazepines).
* BMI more than 40
* Unhealthy dentition.
* Severe bruxers
* TMD patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
The main study parameter/ endpoint is the Apnoea-Hypopnoea Index (AHI) value | from all 6 nights

SECONDARY OUTCOMES:
The secondary study parameter is the Epworth Sleepiness Scale (ESS) | from all 6 nights

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lobbezoo, professor, Study Chair — Academic Centre for Dentistry in Amsterdam
Locations (1):
- Academical Center for dentistry Amsterdam (ACTA), Amsterdam, Netherlands